CLINICAL TRIAL: NCT06512116
Title: An Open Label, Multicenter Phase I Clinical Study Evaluating the Safety, Tolerability, and Pharmacokinetic Characteristics of SIBP-A17 Formulation for Injection in Subjects With Advanced Solid Tumors.
Brief Title: A Clinical Trial of SIBP-A17 Injection in the Treatment of Advanced Solid Tumor Patients.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIBP-A17-I
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor
Keywords: Advanced solid tumor; Her2-ADC; Safety; Efficacy; Pharmacokinetics

STUDY DESIGN:
Intervention Model Description: This study is an open, dose expanding, and indication expanding study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SIBP-A17 (Experimental): SIBP-A17 is an Her2-ADC drug.
  Interventions: Drug: SIBP-A17

INTERVENTIONS:
Drug: SIBP-A17 — Strength: 1, 2, 4, 5, 6 or 8 mg. Intravenous infusion administration, with a treatment cycle of every 21 days, administered once on the first day of each cycle.
  The dose escalation stage, 1mg/kg and 2mg/kg were subjected to accelerated titration, where the safety was evaluated within 21 days after the first administration to one subject. If dose-limiting toxicity (DLT) occurred, the traditional "3+3" dose escalation method was immediately switched. If DLT does not occur, the next dose group will be explored, and the dose exploration starting from 4mg/kg will adopt a "3+3" dose escalation design.
  Other Names: Her2-ADC

SUMMARY:
To evaluate the safety, tolerability, and pharmacokinetic characteristics of SIBP-A17 and determine the maximum tolerable dose (MTD) and phase II recommended dose (RP2D).

DETAILED DESCRIPTION:
This study is an open, dose expanding, and indication expanding study to evaluate the safety, tolerability, pharmacokinetics, immunogenicity, preliminary anti-tumor efficacy, QT/QTc interval effects and explore potential biomarkers of SIBP-A17 in patients with advanced solid tumors.

This study is divided into two stages and is planned to be set up six dose groups, including 1, 2, 4, 5, 6, and 8 mg/kg. The first stage is the dose escalation stage, adopting an improved "3+3" dose escalation design, with a planned enrollment of 14-36 participants. The second stage is the dose expansion stage, where one or two doses are selected to enter the dose expansion phase (4 indication cohorts). 20-40 late-stage solid tumor participants are enrolled in each dose group for dose expansion, and 80-160 participants are planned to be enrolled in the dose expansion phase.

After obtaining certain safety and pharmacokinetic data during the dose escalation phase, the Safety Monitoring Committee (SMC) can discuss and decide whether to synchronize dose expansion.

ELIGIBILITY:
Inclusion Criteria:

* Age range of 18 to 75 years old (including boundary values), gender not limited.
* The clinical diagnosis of enrolled subjects should meet the following criteria:

  1. Dose escalation stage:

     Advanced solid tumor subjects confirmed by histology or cytology to have no standard treatment plan or ineffective or intolerant standard treatment plan.
  2. Dose expansion stage:

     * Cohort 1: Late/unresectable and/or metastatic breast cancer with low HER2 expression (IHC1+or IHC2+/FISH -) after standard treatment failure or intolerance.
     * Cohort 2: HER2 positive (IHC3+or IHC2+and FISH+) local advanced or metastatic digestive system tumors that fail or are not tolerated after standard treatment, including adenocarcinoma of stomach or gastroesophageal junction, colorectal cancer, etc. (pancreatic cancer and biliary tract cancer are excluded).
     * Cohort 3: HER2 positive (IHC3+or IHC2+with FISH+) advanced gynecological tumors that have failed or are intolerant to standard treatment, including but not limited to cervical cancer, endometrial cancer, and ovarian cancer.
     * Cohort 4: Other advanced solid tumors with HER2 expression that failed or were intolerant after standard treatment were preferentially included but not limited to HER2 positive (IHC3+or IHC2+and FISH+) breast cancer (at least 10 cases included), non-small cell lung cancer, etc.
* Willing and able to provide sufficient fresh collected or archived tumor tissue samples (only applicable during dose expansion phase).
* There must be at least one measurable lesion as the target lesion (according to RECIST v1.1 criteria, CT or MRI). Lesions that have received previous radiotherapy or other local treatments are not considered as target lesions unless there is clear progression of the lesion.
* The Eastern Cooperative Oncology Group (ECOG) score for physical fitness is 0 or Expected survival period ≥ 3 months.
* During the screening period, the main organ functions were basically normal [no blood transfusion, granulocyte colony-stimulating factor (G-CSF), or other medical support was received within 14 days before the use of the experimental drug]
* During the screening period, women of childbearing age with negative blood pregnancy test results and reproductive age subjects (including male subjects) who have no pregnancy plans during the trial period and within 6 months after the last dose and voluntarily take effective contraceptive measures.
* Voluntarily participate in this study and sign the informed consent form.

Exclusion Criteria:

* Patients with tumors as specified in the protocol
* Individuals with a history of previous treatment or surgery, or those who have received anti-tumor treatment as specified in the protocol during the planned trial period.
* Individuals with a history of previous illnesses or abnormal conditions as specified in the laboratory examination protocol.
* Screening for individuals with positive Treponema pallidum antibodies during the screening period. Individuals with active hepatitis B virus (HBV) or hepatitis C virus (HCV).
* Patients with ascites, pleural effusion, and pericardial effusion accompanied by clinical symptoms during the screening period who require drainage, or those who have undergone serosal fluid drainage within 4 weeks before the first administration.
* The screening period is accompanied by severe, progressive, or uncontrolled diseases, and it has been assessed by the researchers that participation in the study would increase the risk for the subjects.
* History of interstitial lung disease/non infectious pneumonia in the past, currently suffering from interstitial lung disease/non infectious pneumonia, or suspected interstitial lung disease/non infectious pneumonia that cannot be excluded through imaging examination during screening.
* Subjects who have experienced severe infections within 4 weeks prior to their first medication. Active infections that have received therapeutic intravenous antibiotics within 2 weeks prior to the first medication. Subjects receiving prophylactic antibiotic treatment can be enrolled.
* Participants who have participated in any clinical trial as subjects within the first 3 months of enrollment (excluding subjects who have only participated in clinical trial screening and have not used the investigational drug).
* According to the judgment of the investigator, there are concomitant diseases (such as severe diabetes, thyroid disease, etc.) that seriously endanger the safety of the subject or affect the completion of the study.
* Individuals with a history of severe allergies to protein products, CHO cell products, other recombinant human or humanized antibodies, or components of the investigational drug.
* Pregnant and lactating women.
* Researchers believe that participants who are not suitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Day 126
  During the dose escalation phase, the first treatment cycle (21 days after the first dose) after the subject's administration was determined by the investigator to have occurred events related to the investigational drug as specified in the protocol.
Maximum tolerated dose (MTD) | Day 260
  The maximum tolerated dose (MTD) refers to the highest dose at which DLT does not occur in <1/3 of subjects or ≤ 1/6 of subjects during the DLT observation period.
Recommended Phase II Dose (RP2D) | Day 518
  Recommended Phase II Dose The optimal dose for phase II clinical trial research obtained based on clinical trial results of phase I and literature review.
Adverse Events (AE) | 28 days
  That is adverse events, any adverse events that occurred to the participant during the study period.

SECONDARY OUTCOMES:
AUC (Area Under The Plasma Concentration Versus Time Curve) | 15 days
  It shows the degree to which a drug is absorbed and used in the body.
Cmax (Peak Plasma Concentration) | 15 days
  It shows the highest plasma concentration of a drug that can be achieved after administration.
ORR(Objective Response Rate) | 5 months
  The proportion of participants whose tumor volume shrinks to a predetermined value and maintains the minimum time limit and is the sum of complete and partial responses.
DCR (Disease control rate) | 5 months
  In clinical trials, the percentage of participants with advanced or metastatic cancer who responded fully to cancer treatment, partially responded, and had stable disease.
PFS(Progression-free survival) | 5 months
  The time between the onset of randomization and the onset (of any aspect) of tumor progression or death (from any cause).
OS (overall survival) | 5 months
  From randomization to time of death due to any cause.
Δ QTcF | 15 days
  Changes in Δ QTcF (post administration QTcF baseline QTcF) at various time points after administration.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Huang, Doctor, Principal Investigator — Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical
Locations (1):
- Cancer Hospital of Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No